CLINICAL TRIAL: NCT00498017
Title: Infections After Renal Transplantation: Diseases Pattern in Hong Kong
Status: Completed | Type: Observational
Sponsor: Hospital Authority, Hong Kong (Other Government)
Other Study IDs: KW/EX/06-044; HARECCTR0500060
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Transplantation; Infection
Keywords: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Infections are the most feared complications developing in patient who had had kidney transplantation. The aim of this study is to document the local disease pattern among this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* All living-related or cadaveric renal transplantation episodes (including preemptive ones) performed in the Hong Kong Special Administration Region (HKSAR), Mainland China or overseas during the period 1/1/2000 to 30/6/2005

Exclusion Criteria:

* multiple organ recipients, incomplete records and lost to follow-up, including those cases who have been taken over by other renal centres

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Over a period of 4.5 years, between 1/1/2000 and 30/6/2005, there were totally 58 new cases in our renal transplantation clinic. 36 of them were male, 22 of them were female (Male to female ratio is 1.64:1). All were single-organ recipients. Majority of them (57/58 or 98.3%) were receiving their first renal transplantation, the only exception was a women receiving her second renal transplantation during the study period. Majority (57/48 or 98.3%) of them were cadaveric renal transplantation (CRT). One living-related renal transplantation (LDRT) had been performed in Hong Kong during the study period. Majority of the renal transplantation were performed in Mainland China (48/58 or 82.8%), whilst the remaining 10 operations (17.2%) were performed in Hong Kong.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2006-07; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sze Kit Yuen, Dr, Principal Investigator — Department of Medicine & Geriatrics, ICU, Caritas Medical Centre
Locations (2):
- China (2):
  - Caritas Medical Centre, Hong Kong
  - Princess Margaret Hospital, Hong Kong